CLINICAL TRIAL: NCT02213237
Title: The Application of SERS and Metabolomics in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201107031 RC
Record Dates: First submitted 2013-10-11; First posted 2014-08-11 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It has always been a real challenge to treat sepsis in critically ill patients. The mortality is as high as 20％ in patients with severe sepsis and 46％ with septic shock develops. Early diagnosis and early treatment are the principles. Along with appropriate resuscitation, judicious and thoughtful intravenous antibiotic therapy is the critical determinant of survival in sepsis and septic shock given that ineffective initial therapy worsens the outcome. Blood culture and subsequent susceptibility testing are the gold standard for microbiological diagnosis to direct the optimal use of antibiotic. However, this conventional approach usually takes 5-7 days to wait for the final report. Positive results were reported in only 30% of patients with sepsis and 50 to 60% septic shock. Moreover, the very low bacteria level in blood and prior use of antibiotics may prevent pathogen growth. Surface-enhanced Raman scattering (SERS) is a novel spectroscopy technique based on Raman scattering and localized surface plasma resonance (LSPR), which results in strongly enhanced Raman signals derived from molecules attached to nanometre-sized gold (Au) and silver (Ag) structures. SERS provides the structural information of biomedical molecules with ultra-sensitive characterization down to single molecular level in fast and non-destructive manner. The clinical application of SERS in sepsis will first help to recognize pathogens as well as their specific drug sensitivity, and then optimally guide the initial antibiotics usage. Plasma from twenty blood culture proven Gram positive, negative and Candida cases will separately subject to metabolomics profiling and bioinformatics analysis to establish each pathogen metabolites profile. The sensitivity and specificity of SERS and metabolomics in identifying pathogen and antibiotics-resistant strains will be evaluated. The investigators expected both techniques to play a crucial role in modern sepsis treatment and bring great impact on mortality reduction.

DETAILED DESCRIPTION:
Sepsis is a serious medical condition caused by an overwhelming immune response to infection. Different series of chemicals released into the blood to fight infection trigger systemic inflammation, which is also called systemic inflammatory syndrome, SIRS. Sepsis is one of the major public health issues, which are characterized with high cost and high mortality. Epidemiological studies suggest that there are approximately 300 sepsis cases in per 100,000 population; accounting for 2% of all hospital admissions and up to 30% of intensive care unit admissions. Sepsis is the leading cause of death in critically ill patients. The mortality is as high as 20％ in patients with severe sepsis and 46％ when septic shock develops. Despite recent advances in sepsis treatment, including early goal-directed therapy, low-dose corticosteroid use, protective ventilation, intensive glucose control and activated protein C use, sepsis is still a major challenge for clinical physicians.

Early appropriate antibiotic therapy targeting at the causative pathogen is always crucial to the successful treatment of severe sepsis and septic shock. However, blood culture, the current standard for microbiological diagnosis, can't provide the instant information of pathogens identification at the right beginning of sepsis.

It usually takes 5-7 days to wait for the final report and even much longer for some slow-growth bacteria or yeasts. Moreover, the yield positive rate is low. Only 30% positive results were reported in patients with sepsis and 50 to 60% in septic shock. Some microorganisms are present in the blood in very small numbers and must have longer time to reproduce and grow to quantities that can be detected. Some microorganisms are difficult to grow and special nutrient media may be needed. Viruses cannot be also detected using blood culture bottles designed to grow bacteria. Besides, antimicrobial therapy in the preceding two weeks may prevent pathogen growth.

Since the time to initiation of appropriate antimicrobial therapy is the strongest predictor of mortality, the antibiotics are usually started "empirically" (ie. based on doctors' experience) with broad spectrum and adjusted according to the clinical response. For lack of precise data, inadequate infection control may encounter leading to poor prognosis, and furthermore adverse effects of antibiotics such as organ toxicity and collateral damage (i. e., selection of drug-resistant organisms and the unwanted development of colonization or infection with multidrug-resistant organisms) occurs.

Using the SERS and fluorescent microscopy-based high-speed diagnosis platform for clinical microbiology may help to solve this problem. The specific aims of the subproject are listed as below:

1. To develop a comprehensive protocol of pretreatment of the complex blood sample from the patients with sepsis as the preparation for SERS detection.
2. To identify the causative bacteria or yeasts in the blood by the high-speed diagnosis platform based on SERS to guide the initial antibiotics treatment in sepsis.
3. To examine the susceptibility of the causative pathogen to various antibiotics to guide the initial antibiotics treatment in sepsis.
4. To quantify the bacterial counts in blood to explore the relationship between the load (virulence) of pathogen and clinical course, transmissibility, and antibiotic resistance in patients with sepsis.
5. To compile a database of SERS spectra of clinical microbiology, including bacteria, yeasts and fungi that are the common causative pathogens of sepsis.

The investigators expect this novel technique based on SERS and fluorescent optical microscopy will play a crucial role in modern sepsis treatment, not only bringing great impact on mortality reduction, cost control, but also alleviating the problem of growing resistant trains from the inappropriate use of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

- Any hospitalized patient with

* Septic shock
* Before the use of parenteral or systemic antimicrobial therapy

Exclusion Criteria:

* Pregnant women
* Organ transplantation
* Cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hospitalized patient with Septic shock
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Identification of the causal pathogenic organism of sepsis subjects as well as the drug sensitivity test by SERS technique. | 5-6 hours
  By the SERS technique may measure one time as below:
  1. Reducing detect/diagnosis time of bacteria or yeasts about blood sample of clinical sepsis subjects within one day.
  2. Reducing detect/diagnosis time of bacteria or yeasts for the drug sensitivity test of sepsis subjects within one day.

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Yi Han, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan